CLINICAL TRIAL: NCT04208347
Title: Perioperative Treatment of Combined SOX With Apatinib and Camrelizumab for Resectable Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma: A Multicenter, Randomized Phase II-III Trial
Brief Title: Perioperative Treatment of Combined SOX With Apatinib and Camrelizumab for Oesophagogastric Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRAGON - IV; Ahead-G208 (Other: Ruijin Hospital)
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — apatinib; camrelizumab; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apatinib and Camrelizumab and S-1 and Oxaliplatin (Experimental)
  Interventions: Drug: Apatinib 250mg; Drug: Camrelizumab; Drug: S-1, Oxaliplatin
- Apatinib and S-1 and Oxaliplatin (Experimental)
  Interventions: Drug: S-1, Oxaliplatin; Drug: Apatinib 500mg
- S-1 and Oxaliplatin (Active Comparator)
  Interventions: Drug: S-1, Oxaliplatin

INTERVENTIONS:
Drug: Apatinib 250mg — Apatinib 250mg
  Arms: Apatinib and Camrelizumab and S-1 and Oxaliplatin
Drug: Camrelizumab — Camrelizumab 200mg
  Arms: Apatinib and Camrelizumab and S-1 and Oxaliplatin
Drug: S-1, Oxaliplatin — S-1, Oxaliplatin, q3w
Drug: Apatinib 500mg — Apatinib 500mg
  Arms: Apatinib and S-1 and Oxaliplatin

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of chemotherapy and apatinib with or without camrelizumab in the neoadjuvant (prior to surgery) or adjuvant (after surgery) treatment of previously untreated adults with gastric and gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated localized gastric or GEJ adenocarcinoma as defined by T3-4N+M0;
* Plans to proceed to surgery following pre-operative chemotherapy.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* Has adequate organ function.
* Male participants of childbearing potential must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of therapy.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of therapy.
* Has life expectancy of greater than 12 months.

Exclusion Criteria:

* Uncontrolled hypertension ( systolic ≥140 mmHg or diastolic ≥90 mmHg despite antihypertensive therapy)
* Known hypersensitivity to any of the study drugs or excipients.
* Known hereditary or acquired bleeding and thrombotic tendencies (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, etc.);
* Congenital or acquired immune deficiency (e.g. HIV infected)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Event-free Survival (EFS) | Up to approximately 2 years

SECONDARY OUTCOMES:
Major pathological response(MPR) | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Margin-free (R0) resection rate | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
DFS | up to 2 years
OS | up to 3 years
Downstaging of N stage | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
AEs | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Zhu, Principal Investigator — Ruijin Hospital
Locations (23):
- China (23):
  - Affiliated Hospital of Hebei University, Baoding
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Hainan Cancer Hospital, Haikou
  - Cancer Hospital of the University of Chinese Academy of Sciences, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Hefei Cancer Hospital, Chinese Academy of Sciences, Hefei
  - Lanzhou University Second Hospital, Lanzhou
  - Changhai Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Liaoning Cancer Hospita & Institute, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Jilin Guowen Hospital, Siping
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Tangdu Hospital, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Provincial Cancer Hospital, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang

REFERENCES:
- [Derived] Yang Z, Yu B, Hu J, Jiang L, Jian M. LRRC25 Is a Potential Biomarker for Predicting Immunotherapy Response in Patients with Gastric Cancer. Dig Dis Sci. 2025 Apr;70(4):1395-1410. doi: 10.1007/s10620-025-08882-7. Epub 2025 Feb 17. PMID 39961962
- [Derived] Li C, Tian Y, Zheng Y, Yuan F, Shi Z, Yang L, Chen H, Jiang L, Wang X, Zhao P, Zhang B, Wang Z, Zhao Q, Dong J, Lian C, Xu S, Zhang A, Zheng Z, Wang K, Dang C, Wu D, Chen J, Xue Y, Liang B, Cheng X, Wang Q, Chen L, Xia T, Liu H, Xu D, Zhuang J, Wu T, Zhao X, Wu W, Wang H, Peng J, Hou Z, Zheng R, Chen Y, Yin K, Zhu Z. Pathologic Response of Phase III Study: Perioperative Camrelizumab Plus Rivoceranib and Chemotherapy Versus Chemotherapy for Locally Advanced Gastric Cancer (DRAGON IV/CAP 05). J Clin Oncol. 2025 Feb;43(4):464-474. doi: 10.1200/JCO.24.00795. Epub 2024 Oct 9. PMID 39383487
- [Derived] Zheng Y, Wang Z, Yan C, Yan M, Hou Z, Zheng R, Zhu Z, Li C. Protocol for a randomized controlled trial of perioperative S-1 plus oxaliplatin combined with apatinib and camrelizumab in patients with resectable, locally advanced gastric or gastroesophageal junction adenocarcinoma. Ann Transl Med. 2020 Dec;8(24):1684. doi: 10.21037/atm-20-7802. PMID 33490196
- [Derived] Zheng Y, Yang X, Yan C, Feng R, Sah BK, Yang Z, Zhu Z, Liu W, Xu W, Ni Z, Beeharry MK, Hua Z, Yan M, Zhu Z, Li C. Effect of apatinib plus neoadjuvant chemotherapy followed by resection on pathologic response in patients with locally advanced gastric adenocarcinoma: A single-arm, open-label, phase II trial. Eur J Cancer. 2020 May;130:12-19. doi: 10.1016/j.ejca.2020.02.013. Epub 2020 Mar 11. PMID 32171104